CLINICAL TRIAL: NCT02331498
Title: A Phase I/II Study of Pazopanib in Combination With Temozolomide in Patients With Newly Diagnosed Glioblastoma Multiforme After Surgery and RT-CT
Brief Title: Phase I/II Study of Pazopanib+ Temozolomide in Patients With Newly Diagnosed Glioblastoma Multiforme
Acronym: PAZOGLIO
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Centre Antoine Lacassagne (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012/49
Record Dates: First submitted 2014-11-10; First posted 2015-01-06 (Estimated); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma | interventions — pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A Pazopanib (Other): Open label study with one group
  Interventions: Drug: Pazopanib

INTERVENTIONS:
Drug: Pazopanib — Study drug Pazopanib will be administered once tumoral evaluation has been performed and after Stupp Protocol (TMZ + Radiation) realisation.

SUMMARY:
A phase I/II study of pazopanib in combination with temozolomide in patients with newly diagnosed glioblastoma multiforme after surgery and RT-CT (PAZOGLIO study)

DETAILED DESCRIPTION:
Glioblastoma (GBM), the most common and most malignant primary brain tumor, represents a major medical challenge considering its extremely poor prognosis (Wen 2008). Current standard of care includes maximal surgical resection, followed by concomitant radio-chemotherapy (temozolomide - TMZ) (RT-CT) followed by 6 months of maintenance TMZ, with a median overall survival (mOS) of 14.6 vs. 12.1 months with RT alone (Stupp 2005). Non operable GBM, represents around 30% of cases of GBM, with a poorer prognosis, a median PFS of 3-4 months and a median OS between 6-9 months (Chinot 2007, Stupp 2009), with concomitant RT-CT treatment. Therefore, innovative treatment strategies are urgently needed and new treatment combinations evaluated in phase I studies are highly encouraged (Wen 2011).

Since GBM is one of the most vascularised cancers, antiangiogenic agents have been tested and used firstly in recurrent GBM. Among them, Bevacizumab, a humanized monoclonal antibody against vascular endothelial growth factor (VEGF), has shown high response rate between 19% and 62% in several Phase 2 and multiple retrospective studies, alone or in combination with chemotherapy (Chamberlain 2011). Two randomized phase III trials, AVAGLIO and RTOG 0825, investigating the efficacy of Bevacizumab added or not to the Stupp protocol in patients with newly diagnosed GBM, have been presented at the annual meeting of the American Society of Clinical Oncology (ASCO 2013). While both studies exhibited a significant progression-free survival (PFS) improvement (RTOG 0825:10.7 vs. 7.3m, p=0.007; AVAGLIO: 10.6 vs. 6.2m, p<0.0001), there was no gain in overall survival.

Other antiangiogenic agents have been studied in GBM patients (Sathornsumetee 2009, Van Meir 2010, Wick 2011), with encouraging results but still insufficient when used as single agents. Among them, pazopanib is thought to be promising. It is an orally tyrosine kinase inhibitor with potently inhibition of VEGFR-1, -2, -3, c-kit and PDGFR-α, -β (Castaneda 2009, Schutz 2011). Interestingly, these 2 PDGFR subtypes are overexpressed in malignant gliomas (Verhaak 2010). Furthermore, pazopanib is already validated in patients with advanced renal cell carcinoma and soft-tissue sarcomas (Sleijfer 2009, Sternberg 2010).

A phase II trial evaluated efficacy and safety of pazopanib in 35 patients with recurrent GBM (Iwamoto 2010). Two patients had a partial radiographic response by standard bidimensional measurements, whereas 9 patients (6 at the 8-week point and 3 only within the first month of treatment) had decreased contrast enhancement, vasogenic edema, and mass effect but <50% reduction in tumor. The median PFS was 12 weeks and mOS was 35 weeks. Pazopanib was reasonably well tolerated with a spectrum of toxicities similar to other anti-VEGF/VEGFR agents and with unexpected toxicity.

Given the emerging concern that pure anti-VEGF inhibition may promote malignant glial cell invasiveness (Keunen 2011), we consider essential to combine a multitargeted antiangiogenic agent, such as pazopanib, with the current standard treatment. TMZ was chosen not only because it represents the current standard of care but because of its very good penetration in the brain parenchyma and its low hepatic metabolism, making very unlikely the occurrence of a pharmacokinetic interaction with pazopanib (Friedman 2000). Indeed, phase I trials of TMZ in combination with molecules such as RAD001, cilengitide, gefitinib or irinotecan showed no need for dose modification of TMZ. Similarly, the Phase I trials of pazopanib association with paclitaxel or FOLFOX6 have been conducted up to a dose of 800 mg daily, the recommended dose of pazopanib in monotherapy, with standard doses of chemotherapy (Tan 2010, Brady 2009). Finally, the study of the toxicity profile of pazopanib and TMZ does not suggest a specific limiting dose escalation adverse event, except perhaps asthenia, thrombocytopenia or ALAT elevation. However, considering the high level of potential toxicity when an ITK is administered with radiations, pazopanib should not be administered in the induction phase of the Stupp protocol.

Therefore, based on a strong synergy rational, the study coordinator aims to evaluate the safety and efficacy of pazopanib in combination with TMZ in the maintenance phase of the Stupp protocol. The study coordinator hopes that this strategy could significantly improve the poor prognosis of these patients.

This study is a multicenter Phase I/II trial, which aims to determine the Recommended Phase 2 Dose (RP2D) of pazopanib in combination with TMZ. The study coordinator will associate a multidisciplinary approach involving translational pharmacokinetic studies, and research on potential predictive biomarkers of response through pharmacogenetic and pharmacogenomic approachs. This study will include patients with not previously treated GBM, candidates for a complete or partial surgical resection and who are eligible for adjuvant treatment based on a combination of TMZ and radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must provide written informed consent prior to performance of study-specific procedures or assessments and must be willing to comply with treatment and follow up.
* Age ≥ 18 years and < 70 years
* Histologically confirmed diagnosis of GBM
* Surgically treated other than exclusive biopsy (complete or partial resection) of the GBM, for which adjuvant radiotherapy and chemotherapy is indicated
* Eligibility criteria that will need to be checked before patient registration and - No TMZ interruption resulting in hematological toxicity should has occurred
* AND the delivery of radiation dose as defined in the Stupp protocol should be at least equal to 80%
* Eastern Cooperative Oncology Group (ECOG) performance status of Glioblastoma ≤ 2
* Life expectancy>3 months
* Measurable disease criteria : Based on the RANO criteria (Wen 2010) objective tumor response will be assessed by MRI and 18F-DOPA PET)
* Archived tumor tissue must be available for all subjects for biomarker analysis before and/or during treatment with investigational product.
* Stable doses of corticosteroid for more than 1 week.
* Adequate biological function
* Women of childbearing potential must have a negative serum pregnancy test within 14 days of first dose of study treatment and agree to use effective contraception, as defined in Pregnancy Section in overall Safety Section during the study and for 6 months following the last dose of investigational product.

Exclusion Criteria:

* Prior malignancy.
* Surgical treatment consisting in exclusive biopsy or absence of initial surgery
* Pre-treated GBM
* Allergy to any of the tested drugs
* Clinically significant gastrointestinal abnormalities that may increase the risk for gastrointestinal bleeding including,
* Clinically significant gastrointestinal abnormalities that may affect absorption of investigational product
* Corrected QT interval (QTc) > 480 msecs
* History of any one or more of ardiovascular conditions within the past 6 months
* Poorly controlled hypertension
* History of cerebrovascular accident including transient ischemic attack (TIA), pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months.
* Major surgery or trauma within 28 days prior to first dose of investigational product and/or presence of any non-healing wound, fracture, or ulcer (procedures such as catheter placement not considered to be major surgery).
* Evidence of active bleeding or bleeding diathesis.
* Known endobronchial lesions and/or lesions infiltrating major pulmonary vessels that increase the risk of pulmonary hemorrhage
* Recent hemoptysis
* Any serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with subject's safety, provision of informed consent, or compliance to study procedures.
* Unable or unwilling to discontinue use of prohibited medications listed in Appendix C for at least 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of study drug and for the duration of the study (Appendix C).
* Treatment with any of the following anti-cancer therapies:

  * radiation therapy, surgery or tumor embolization within 14 days prior to the first dose of pazoapnib OR
  * chemotherapy, immunotherapy, biologic therapy, investigational therapy or hormonal therapy within 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of Pazopanib
* Administration of any non-oncologic investigational drug within 30 days or 5 half-lives whichever is longer prior to receiving the first dose of study treatment
* Any ongoing toxicity from prior anti-cancer therapy that is >Grade 1 and/or that is progressing in severity, except alopecia.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2015-06 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
Recommended Phase 2 Dose (RP2D) of pazopanib in oral route in addition to the maintenance phase of the Stupp protocol, according the rate (33 %) of tolerate toxicities | phase I
  To evaluate the Recommended Phase 2 Dose (RP2D) of pazopanib in oral route in addition to the maintenance phase of the Stupp protocol, regarding the toxicities that should not be more than 33 %

SECONDARY OUTCOMES:
overall tolerance of pazopanib : number of biological toxicities, blood pressure and hemorragic events | 2 years
  To define the overall tolerance of pazopanib associated with TMZ during the maintenance phase of the "Stupp protocol" regarding biological toxicities, blood pressure and hemorragic events
antitumor activity of the adjunction of daily dose of pazopanib to the maintenance phase of the Stupp protocol | 2 years
  To assess the antitumor activity of the adjunction of daily dose of pazopanib to the maintenance phase of the Stupp protocol according to the Revised Assessment in Neuro-Oncology (RANO) criteria (response rate) and the median duration of response.
determine the median Progression-Free-Survival | 12 months
  To determine the median Progression-Free-Survival (mPFS), the PFS rate at 12 (PFS-12) months.
determine the median Overall Survival (mOS) | 12 months
  To determine the median Overall Survival (mOS), the OS rate at 6 (OS-6) and 12 (OS-12) months.
pharmacokinetics profile: area under curve regarding plasma concentration /time between 0 and 8 h (AUC0-8 hours) from 0 to 24 h (AUC 0-24 hours), maximum plasma concentration (Cmax), time to the concentration maximum (Tmax) and plasma half-life (t1/2) | 2 years
  To determine the pharmacokinetics (PK) profile of pazopanib when given in combination with TMZ.
determine the pharmacokinetics (PK) profile of TMZ | 2 years
  To determine the pharmacokinetics (PK) profile of TMZ when given in combination with pazopanib.

CONTACTS AND LOCATIONS:
Overall Officials: Christine LOVERA, Study Director — Centre Antoine Lacassagne
Locations (1):
- Centre Antoine Lacassagne, Nice, Cedex 2, France

REFERENCES:
- See also: website — http://www.centreantoinelacassagne.org